CLINICAL TRIAL: NCT06206252
Title: The Effect of Medical Cannabis on Opioid Use for Individuals with Chronic Pain
Brief Title: Can Medical Cannabis Affect Opioid Use?
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: iRIS-2022-1273
Record Dates: First submitted 2023-06-15; First posted 2024-01-16 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain; Pain
Keywords: Prescription opioids; Medical Cannabis
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Medical Cannabis Group: Participants will use designated medical cannabis products for the study duration.
  Interventions: Other: Medical Cannabis
- Control Group: Participants will not use any cannabis for the study duration.

INTERVENTIONS:
Other: Medical Cannabis — Participants will be restricted to specific medical cannabis products from Ethos Dispensary. They will be randomized to one medical cannabis formulation (tincture or vaporization) for the duration of the study. Each month for three months, they will purchase a different composition (predominantly THC, predominantly CBD, or balanced products) of their designated formulation. The order of compositions will be randomized and double-blinded, so participants and the research team will not know which compositions of medical cannabis they are using each month.
  Groups: Medical Cannabis Group

SUMMARY:
The goal of this observational study is to learn how medical cannabis (MC) affects pain and the use of opioid pain medications. Participants who have chronic pain and use prescribed opioid pain medication will opt-in to using MC or not for the 3-month study. Participants who are certified in Pennsylvania will purchase specific medical cannabis products at a reduced cost from a partnering medical cannabis dispensary monthly. All participants will complete baseline, daily, and monthly assessments to observe changes across groups.

DETAILED DESCRIPTION:
The primary aim is to observe if individuals who have chronic pain that they are treating with opioids and medical cannabis report changes in pain severity, function, and opioid use compared to those who do not use medical cannabis.

Secondary aims include observation of whether the use of medical cannabis differentially impacts tolerability (side effects, risk of cannabis use disorder), sleep-related symptoms, or quality of life and mental health among chronic opioid users.

There will be two groups, participants who are certified to use medical cannabis and those who do not use any cannabis. All participants will complete a baseline survey to report demographics, pain, sleep, mental health, well-being, quality of life, and use of medications. Some of these questions will be repeated monthly. Participants will also receive a link via text to a daily survey to report daily prescription opioid use and medical cannabis use (if applicable) as well as pain severity and interference.

Participants who purchase medical cannabis at Ethos will be randomized and restricted to one formulation of medical cannabis (vaporization or tincture) for the study duration. They will purchase three different compositions of the specific medical cannabis formulation at a reduced cost over 3 months and the order of those compositions will be randomized. They will purchase one composition per month and they will not know which one they are purchasing. The three different compositions are:

* A composition that is predominantly THC (tetrahydrocannabinol)
* A composition that is predominantly CBD (Cannabidiol)
* A composition that is a one-to-one blend of THC and CBD

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of chronic, intractable pain
* Use of prescription opioids for longer than 90 days
* Have a smartphone or agree to use one provided
* English fluency
* Medical cannabis group only: Willing to get certified by a physician to use medical cannabis in PA OR already certified but have not been using medical cannabis products regularly (daily or weekly) for longer than 30 days
* Medical cannabis group only: Willing to accept a temporary restriction on medical cannabis products
* Control group: Agree to continue not using cannabis for the duration of the study (3 months)

Exclusion Criteria:

* Under 18 years old
* Being under conservatorship
* Self-reported pregnant or breastfeeding
* Cannabis Use Disorder
* Active treatment in methadone or buprenorphine program for Opioid Use Disorder
* Diabetic neuropathy or chemotherapy-induced neuropathy alone
* Medical cannabis group: Cannabis use (daily/weekly) for more than 30 days
* Control group: Cannabis Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 110 individuals with chronic pain who use prescribed opioids (90 medical cannabis users, 20 non-users) and live in Pennsylvania will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity | Baseline, 4 weeks, 8 weeks, 12 weeks
  Measured using Brief Pain Inventory Short Form (BPI-SF), scores 0-10 with higher scores indicating more pain severity
Change in pain interference | Baseline, 4 weeks, 8 weeks, 12 weeks
  Assessed using Brief Pain Inventory Short Form (BPI-SF), scores 0-10 with higher scores indicating more pain interference
Change in pain | Daily up to 12 weeks
  Assessed using Pain, Enjoyment of Life and General Activity Scale (PEG Scale), scores 0-10 with higher scores indicating more pain
Change in daily use of prescription opioids | Daily up to 12 weeks
  Assessed using self-reported number of prescription opioids taken in last 24 hours

SECONDARY OUTCOMES:
Change in quality of life | Baseline, 4 weeks, 8 weeks, 12 weeks
  Assessed using Linear Analog Scale Assessment, scores 0-10, higher scores indicating better quality of life
Change in mental health status | Baseline, 4 weeks, 8 weeks, 12 weeks
  Assessed using Patient Health Questionnaire-4 (PHQ-4), scores 0-12, higher scores indicating severe anxiety and depression
Change in sleep quality | Baseline, 4 weeks, 8 weeks, 12 weeks
  Assessed using Insomnia Severity Index (ISI), scores 0-28, higher scores indicating more severe insomnia
Side effects of medical cannabis | Baseline, 4 weeks, 8 weeks, 12 weeks
  Assessed using sum of side effects self-reported, higher scores indicating higher rates of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Worster, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided